CLINICAL TRIAL: NCT07266974
Title: Evaluation of Post -Operative Pain After Obturation Using Two Different Types of Sealers - A Randomized Clinical Trial
Brief Title: To Evaluate Post Operative Pain Using Two Different Kind of Sealers in Obturation of Teeth With Symptomatic Irreversible Pulpitis During Second Visit When the Patient is Painless
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jaweria Gul Keyani (Other)
Responsible Party: Sponsor-Investigator, Jaweria Gul Keyani, Post Graduate Trainee, Margalla Institute of Health Sciences
Organization: Margalla Institute of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DJ/277/25
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Post Operative Pain, Acute; Irreversible Pulpitis
Keywords: post operative pain; bioceramic sealer; irreversible pulpitis
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A , AH plus sealer , Group B ( bioceramic sealer) (Active Comparator): patients in group A will recieve AH plus sealer and in group B shall recieve bioceramic sealer for obturation during root canal treatment
  Interventions: Drug: bioceramic sealer
- Group A , (AH plus sealer ) , Group B ( bioceramic sealer) (Active Comparator): patients in Group A will recieve Ah plus sealer for obturation and patients in group B shall recieve bioceramic sealer for obtration during root canal treatment second visit
  Interventions: Drug: AH-Plus Epoxy Resin Sealer

INTERVENTIONS:
Drug: AH-Plus Epoxy Resin Sealer — AH plus sealer is an epoxy resin based sealer that is biocompatible with good sealing ability
  Arms: Group A , (AH plus sealer ) , Group B ( bioceramic sealer)
Drug: bioceramic sealer — MTA based sealers,biocermic sealers are biocompatible, safe to use
  Arms: Group A , AH plus sealer , Group B ( bioceramic sealer)

SUMMARY:
The goal of this randomized clinical trial is to evaluate pain after root canal treatment using two different kinds of sealers during obturation in 60 healthy , male and female patients ages between 18 to 40 years. The main aims is to systematically evaluate and compare post-operative pain levels in patients undergoing root canal treatment with two different types of endodontic sealers: AH plus (SEAL APEX) and bio ceramic sealer(META)

• By identifying the sealer that leads to the least discomfort, this research could significantly enhance patient care, minimize recovery time, and improve overall treatment success in endodontics.

Participants in both groups will be given a visual analogue scale(VAS) to measure the pain level after the root canal treatment has been completed. They will measure pain levels at 12, 24 and 48 hours. All information will be recorded on proforma and compared.

DETAILED DESCRIPTION:
•This randomized clinical trial is done to evaluate and compare post operative pain after obturation using two different sealers .A total of 60 participants will be selected using a non-probability consecutive sampling method. After enrollment, participants will be randomly allocated into two equal groups (30 each),Group A and Group B using the lottery method. Group A patients will be given AH plus sealer and Group B will be given bio-ceramic sealer. Root canal treatment will be performed in two visits using local anesthesia under rubber dam isolation. • After drying with paper points , in group 1 an even ratio of 1:1 from the base and catalyst of the AH plus will be manually mixed on a paper pad with a spatula and introduced into the canal on the master cone.

* In group B, sealer will be introduced with the bio ceramic sealer tube and cold lateral compaction technique will be used for obturation in both of the groups . Composite will be used for restoration.
* The patients will be called again for evaluation of pain and its severity at, 24hrs, 48hrs and 72hrs. Effectiveness of sealers will be measured as no, mild, moderate or severe pain on visual analogue scale (VAS). All procedures will be done under the supervision of supervisor. All this information will be recorded on proforma.
* Patients shall be prescribed ibuprofen 400mg post-operatively shall be prescribed. Patients will be given VAS scale so they can record their pain at home before taking the analgesic.
* Data will be entered and analyzed in IMB SPSS version 26. Mean and Standard deviation (SD) of VAS scores at each time point (12h, 24h, 48h) for both types of sealers shall be calculated. Independent t-test to compare the VAS scores between two groups (Sealer 1 vs. Sealer 2).
* Significance level to set at p value <0.05 this study will further add to the literature regarding the efficacy of sealer in reducing post operative pain and assessing which sealer is better and effective to use for clinicians.

ELIGIBILITY:
Inclusion Criteria:

* • Patients ranging from 18 to 40 years.

  * Patients whose teeth have been diagnosed with Symptomatic irreversible pulpitis.
  * maxillary and mandibular teeth.
  * A normal periapical condition on radiograph, or one with little to no periodontal ligament (PDL) space widening, confirming the normal periapical state.
  * Teeth that can be restored.
  * Teeth with healthy periodontium.

Exclusion Criteria:

* Non-restorable teeth.
* Patients with poor health whose systemic complications could change the course of treatment.
* Teeth with immature roots.
* Teeth with periapical lesions or apical periodontitis.
* Teeth with Necrotic pulp.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
post operative pain in both sealer groups after obturation | 6 months
  Post-operative pain levels will be measured and compared in both groups using Visual Analogue Scale (VAS) Patients were asked to rate their pain on a numerical scale from 0 to 10, where 0 indicated no pain and 10 indicated the worst pain imaginable.
  For interpretation, pain intensity was categorized as follows:
  1-3: Mild pain
  4-6: Moderate pain
  7-10: Severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Margalla Institute of Health Sciences, Gulraiz phase III Quaid e azam Avenue, Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No